CLINICAL TRIAL: NCT04525417
Title: Use of Rapid Covid-19 Antibody Test Marketed by AAZ Laboratories in Healthcare Workers Presumably Being Infected by SARS-CoV-2
Brief Title: Rapid Screening Test for Covid-19 Antibodies in Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe d'Etude sur le Risque d'Exposition des Soignants aux Agents Infectieux (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GERES20200409; ID RCB 2020-A01031-38 (Other: ANSM)
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-08

CONDITIONS: Covid-19 Immune Status of Healthcare Workers

STUDY DESIGN:
Intervention Model Description: Monocentric, open-label, prospective, non-randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hospital healthcare workers (Other): Clinical examination; Veinous blood sampling for serological testing; capillary drawing to perform a rapid Covid-19 test
  Interventions: Diagnostic Test: AAZ Covid-19 rapid test
- private health professionals (Other): Clinical examination; Veinous blood sampling for serological testing; capillary drawing to perform a rapid Covid-19 test
  Interventions: Diagnostic Test: AAZ Covid-19 rapid test

INTERVENTIONS:
Diagnostic Test: AAZ Covid-19 rapid test — To assess the immune status
  Other Names: ELISA test

SUMMARY:
The study objectives were to assess 1/the immune status of healthcare professionals with suggestive symptomatology of Covid-19 infection and 2/the sensitivity and specificity of AAZ rapid test by comparing it with a serological ELISA test.

An open-label, monocentric, prospective, non-randomized study, is conducted, including 50 hospital healthcare professionals and 50 private health professionals.

Knowledge of serostatus will achieve the implementation of a strategy of management of patients according to specific immunity of health professionals

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals with symptoms suggestive of Covid-19 infection

Exclusion Criteria:

* any other subject
* pregnant women
* protected adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
To assess the predictive value of Covid-19 rapid test | One week
  Comparative study with Elisa Test
Compare the results of rapid tests on serum and capillary samples | one week
  Performance evaluation of rapid tests according to the samples used

SECONDARY OUTCOMES:
A posteriori diagnosis of a covid-19 recent infection with suggestive symptomatology | one week
  Use of rapid test
Analysis of factors associated with negativity of PCR test on oropharyngeal swabs and positive serology | One week
  Analysis of clinical data

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Bouvet, MD, Principal Investigator — Groupe d'Etude sur le Risque d'Exposition des Soignants aux Agents Infectieux
Locations (1):
- Bichat University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No